CLINICAL TRIAL: NCT03626714
Title: An Open-Label, First-in-human, Safety and Pharmacokinetic Study of 1-Month Sustained-Release Injectable Tacrolimus in Healthy Subjects
Brief Title: Safety and Pharmacokinetics of Sustained-release Depot Tacrolimus: A First-in-human Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Auritec Pharmaceuticals (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTB-010; U44AI069674 (NIH)
Record Dates: First submitted 2018-07-31; First posted 2018-08-13 (Actual); Results first posted 2019-06-11 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-07

CONDITIONS: Organ Transplant Rejection; Psoriasis
Keywords: Tacrolimus; Immunosuppressant; Sustained-release; Plexis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sustained Release Tacrolimus (Experimental): All subjects will be treated with a single dose injection of sustained-release Tacrolimus
  Interventions: Drug: Sustained Release Injectable Tacrolimus

INTERVENTIONS:
Drug: Sustained Release Injectable Tacrolimus — Long-acting formulation of tacrolimus developed using Auritec's proprietary Plexis drug delivery technology.

SUMMARY:
This first-in-human study is designed to assess the safety and pharmacokinetic (PK) profile of sustained-release (SR) depot tacrolimus, which will be administered as a single dose of 0.1 mg/kg by subcutaneous (SC) injection in healthy subjects.

DETAILED DESCRIPTION:
This is a first-in-human study to assess the safety and pharmacokinetic (PK) profile of sustained-release (SR) tacrolimus, which will be administered as a single dose of 0.1 mg/kg by subcutaneous (SC) injection in healthy subjects.

The short-term general investigational plan is to evaluate sustained release tacrolimus in healthy volunteers for up to 30 days in an exploratory trial to determine safety and drug concentrations in blood. The results from this study will inform the long-term goal of this program, which is to provide an improved treatment modality for prophylaxis of organ (kidney, liver and heart) transplant rejection with the additional benefit of enhancing medication compliance. These improvements have the potential to mitigate both the personal and economic burden of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to understand and provide informed consent. A signed informed consent form must be provided before any study assessments are done;
* Males or females, between 18 and 45 years of age, inclusive;
* Body mass index must be within the range 18.5 to 32.0 kg/m2, inclusive;
* Must be in good health, as determined by no clinically significant findings from medical history, vital signs, and 12-lead electrocardiogram (ECG), inclusive of documented absence of QT prolongation;
* Clinical laboratory evaluations (including clinical chemistry panel [fasted at least 10 hours], complete blood count [CBC], and urinalysis [UA]) must be within the reference range for the test laboratory, unless deemed not clinically significant by the Investigator;
* Must be negative for autoimmune disorders in the past 3 months and at Screening - participant's medical history will be used for this evaluation;
* Must not use any immunosuppressant calcineurin inhibitor product other than SR Injectable tacrolimus throughout the dosing period and until after the final visit;
* Must agree to blood draws throughout the course of the study and venous access sufficient to allow for blood sampling as per the protocol;
* Must be negative for selected drugs of abuse at Screening and at Check-in (Day -1);
* Must have a negative hepatitis panel (including hepatitis B surface antigen [HBsAg] and hepatitis C virus antibody [HCV]) and negative human immunodeficiency virus [HIV] antibody screens;
* Females will be nonpregnant, nonlactating, and either postmenopausal, defined as amenorrhea for at least 1 year and follicle-stimulating hormone levels of 40 mIU/mL or higher; surgically sterile (eg, tubal ligation, hysterectomy, oophorectomy) for at least 90 days prior to Screening; or agree to use, from the time of signing the informed consent or 10 days prior to Check-in on Day -1 of the Inpatient Period until 30 days after Study Discharge, one of the following forms of contraception: nonhormonal intrauterine device (IUD) with spermicide; female condom with spermicide; contraceptive sponge with spermicide; diaphragm with spermicide; cervical cap with spermicide; male sexual partner who agrees to use a male condom with spermicide; or sterile sexual partner; alternatively, women must agree to maintain abstinence (must agree to use a double barrier method if they become sexually active during the study. For all females of childbearing potential, the pregnancy test result must be negative at Screening and Check-in on Day -1 of the Inpatient Period (see Appendix 1). Women must also agree not to douche throughout the dosing period and until after the final visit;
* Males will either be sterile or agree to use, from Check-in on Day -1 of the Inpatient Period until 90 days following Study Discharge, one of the following approved methods of contraception: male condom with spermicide; sterile sexual partner; or use by female sexual partner of an IUD with spermicide; a female condom with spermicide; a contraceptive sponge with spermicide; an intravaginal system (eg, NuvaRing®); a diaphragm with spermicide; a cervical cap with spermicide; or oral, implantable, transdermal, or injectable contraceptives. Subjects will refrain from sperm donation from Check-in on Day -1 of the Inpatient Period until 90 days following Study Discharge.

Exclusion Criteria:

* Inability or unwillingness of a participant to give written informed consent or comply with study protocol;
* Prisoners or patients who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (eg, infectious disease) illness must not be enrolled into this trial;
* Presence of an uncontrolled, unstable clinically significant medical condition that in the opinion of the Investigator may increase the risk to the subject or may interfere with the interpretation of safety and PK evaluations, or could impair the subject's ability to complete the trial, or could impair the decisional capacity of the subject;
* Presence of clinically significant vital signs or a physical examination finding that, in the opinion of the Investigator, could increase the risk to the subject or may potentially interfere with the ability to evaluate safety and tolerability in the trial;
* History of tacrolimus use, or hypersensitivity and/or adverse reaction to calcineurin inhibitor drugs;
* History of toxic shock syndrome;
* Currently receiving chemotherapy or immunosuppressive agents;
* Use of investigative drugs within 30 days or 5 half-lives of study participation;
* Currently using sirolimus;
* Currently using live vaccines;
* Currently on concomitant substrates and/or inhibitors of CYP3A4;
* Requires the use of any concomitant medication, except for treatment of an adverse event (AE) during the study;
* Any abnormality on clinical laboratory tests, or ECG finding that is considered to be clinically significant by the Investigator.
* Known or suspected (nonfebrile) seizure disorder;
* Use of any other depot medications within the last three months.
* Unwilling to commit to avoid eating grapefruit or drinking grapefruit juice during the first 30 days of this exploratory study.
* Grade ≥ 1 finding as described in the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-01-05 (Actual); Study Completion 2019-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George J Atiee, MD, Principal Investigator — Worldwide Clinical Trials
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Sustained Release Injectable Tacrolimus: All subjects will be treated with a single dose injection of sustained-release Tacrolimus.
Period: Overall Study
Arm/Group | Experimental: Sustained Release Injectable Tacrolimus
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental: Sustained Release Injectable Tacrolimus
Number analyzed (Participants) | 8
Age, Continuous [Mean (Full Range); unit: years] | 34.37 [22 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects That Experienced Treatment-related Adverse Events [Safety and Tolerability]
Description: Adverse events were documented at each study visit according to the criteria set forth in the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials as follows:
  Grade 1 (mild); Grade 2 (moderate); Grade 3 (severe); Grade 4 (potentially life-threatening).
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Groups:
- Experimental: Sustained Release Injectable Tacrolimus: All subjects were subcutaneously injected a single dose (0.1 mg/kg) of sustained-release tacrolimus.
Arm/Group | Experimental: Sustained Release Injectable Tacrolimus
Number analyzed (Participants) | 8
Participants
  Tenderness at Injection Site - Grade 1 | 6
  Burning Pain at Injection Site - Grade 1 | 6
  Erythema/Redness at Injection Site - Grade 1 | 3
  Induration/Swelling at Injection Site - Grade 1 | 2
  Tenderness at Injection Site - Grade 2 | 1

2. Primary Outcome: Drug Concentrations in Blood Samples at Individual Time-points
Description: The concentrations of tacrolimus in blood samples were measured at baseline, day 1 (1 hr, 3 hrs, 6 hrs, 12 hrs, and 24 hrs), followed by days 3, 7, 14, 21, 30, 37, 44, 51 and 60.
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Experimental: Sustained Release Injectable Tacrolimus
Number analyzed (Participants) | 8
ng/mL
  Baseline | 0 (0)
  Day 1, hour 1 | 0.667 (0.505)
  Day 1, hour 3 | 0.956 (0.556)
  Day 1 hour 6 | 1.30 (0.623)
  Day 1, hour 12 | 1.84 (0.548)
  Day 1, hour 24 | 1.54 (0.484)
  Day 3 | 1.24 (0.397)
  Day 7 | 0.775 (0.365)
  Day 14 | 0.341 (0.158)
  Day 21 | 0.320 (0.127)
  Day 30 | 0.302 (0.091)
  Day 37 | 0.282 (0.074)
  Day 44 | 0.260 (0.082)
  Day 51 | 0.269 (0.091)
  Day 60 | 0.260 (0.072)

3. Primary Outcome: Mean Blood Concentration-time Curve - Cmax
Description: Maximum observed tacrolimus whole blood concentration
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Experimental: Sustained Release Injectable Tacrolimus
Number analyzed (Participants) | 8
ng/mL | 1.92 (0.527)

4. Primary Outcome: Mean Blood Concentration-time Curve - Tmax
Description: Time to maximum observed tacrolimus whole blood concentration
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Experimental: Sustained Release Injectable Tacrolimus
Number analyzed (Participants) | 8
Hour | 14.3 (6.36)

5. Primary Outcome: Blood Concentration-time Curve [AUC]
Description: Area under the concentration-time curve
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | Experimental: Sustained Release Injectable Tacrolimus
Number analyzed (Participants) | 8
hour*ng/mL | 568 (171)

6. Primary Outcome: Terminal Elimination Half-life [t1/2]
Description: The apparent terminal elimination half-life was calculated.
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Experimental: Sustained Release Injectable Tacrolimus
Number analyzed (Participants) | 8
hours | 1100 (803)

ADVERSE EVENTS:
Time Frame: For this single-dose experimental study, adverse event data was collected from subjects for up to 60 days.
Arm/Group | Experimental: Sustained Release Injectable Tacrolimus
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Sustained Release Injectable Tacrolimus (N=8)
Elevated Bilirubin (Blood and lymphatic system disorders) | 2
Decreased Hemoglobin (Blood and lymphatic system disorders) | 3
Decreased Platelets (Blood and lymphatic system disorders) | 1
Elevated Alt/Ast (Gastrointestinal disorders) | 1
Elevated Aspartate (Gastrointestinal disorders) | 3
Hypercalcemia (Blood and lymphatic system disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hyperglycemia (General disorders) | 3
Hypoglycemia (General disorders) | 1
Hypokalemia (Renal and urinary disorders) | 1
Hyponatremia (Blood and lymphatic system disorders) | 1
Bruising (General disorders) | 1
Odontalgia left upper wisdom tooth (Musculoskeletal and connective tissue disorders) | 1

LIMITATIONS AND CAVEATS:
The study's main limitations include the small sample size (n=8) and the short duration (60 days).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/14/NCT03626714/Prot_SAP_000.pdf